CLINICAL TRIAL: NCT02175693
Title: Post-marketing Surveillance of Administration of Botulinum Toxin Type B(NerBloc)-Investigation of the Clinical Condition and Safety in Patients With Cervical Dystonia
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: NB01S
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2018-03

CONDITIONS: Cervical Dystonia
Keywords: Torticollis; rimabotulinumtoxinB
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- E2014

SUMMARY:
Investigation of the clinical condition and safety in patients with cervical dystonia

ELIGIBILITY:
Inclusion criteria:

Patients with cervical dystonia

Exclusion criteria:

The patients who participated in this surveillance in the past

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cervical dystonia
Sampling Method: Non-Probability Sample
Enrollment: 1647 (Actual)
Dates: Start 2013-04-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Overall assessments of the improvement in the seriousness of seizures | Up to 3 years
  Improvement is based on the 5 following elements: 1) Eminent improvement 2) Improvement 3) Improvement a little invariability 5) Exacerbation 6) It is not possible to judge

CONTACTS AND LOCATIONS:
Overall Officials: Akira Endo, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo